CLINICAL TRIAL: NCT00143754
Title: Benefit of Controlled Rehydration in Unexplained Syncope
Brief Title: Effect of Chronic Oral Hydration in Patients With Recurrent Unexplained Syncope
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CP00-02; Centre Evian pour l'Eau
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2005-09-02 (Estimated); Status verified 2005-08

CONDITIONS: Hydration; Loss of Consciousness; Neurocardiogenic Syncope
MeSH Terms: conditions — Unconsciousness; Syncope, Vasovagal

INTERVENTIONS:
Procedure: Hydration

SUMMARY:
Beneficial effect of chronic hydration with salt supplementation in patients with recurrent unexplained syncope is not established. We sought to determine if chronic oral rehydration with salt supplementation improved the tolerance and hemodynamic responses of patients with unexplained recurrent syncope.

ELIGIBILITY:
Inclusion Criteria:

* Syncopal and/or near syncopal episodes at least twice within the prior 3 months

Exclusion Criteria:

* Neurological disease
* Structural heart disease
* Metabolic and psychiatric illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Georges PN Leftheriotis, MD-PhD, Principal Investigator — HUAngers